CLINICAL TRIAL: NCT05765253
Title: A Prospective, Multicenter, Randomized Study Evaluating Portal Vein Access Sets During Transjugular Intrahepatic Portosystemic Shunt (TIPS) Procedures
Brief Title: Achieving Portal Access With Scorpion Post-Approval Study (APASS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low patient accrual
Sponsor: Argon Medical Devices (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCPVA01
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Portal Hypertension; Liver Diseases; Ascites Hepatic; Hydrothorax; Vascular Diseases
Keywords: Transjugular Intrahepatic Portosystemic Shunt; TIPS; Portal Vein Access
MeSH Terms: conditions — Hypertension, Portal; Liver Diseases; Hydrothorax; Vascular Diseases | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TIPS with Scorpion Portal Vein Access Kit (Active Comparator): Scorpion or Scorpion X access set
  Interventions: Device: Scorpion Portal Vein Access Kit; Procedure: Transjugular Intrahepatic Portosystemic Shunt (TIPS)
- TIPS with Cook Transjugular Liver Access Set (Active Comparator): Ring or Rosch-Uchida access set
  Interventions: Device: Cook Transjugular Liver Access Set; Procedure: Transjugular Intrahepatic Portosystemic Shunt (TIPS)

INTERVENTIONS:
Device: Scorpion Portal Vein Access Kit — Portal Vein Access with Scorpion or Scorpion X set
  Arms: TIPS with Scorpion Portal Vein Access Kit
Device: Cook Transjugular Liver Access Set — Portal Vein Access with Ring or Rosch-Uchida set
  Arms: TIPS with Cook Transjugular Liver Access Set
Procedure: Transjugular Intrahepatic Portosystemic Shunt (TIPS) — Transjugular Intrahepatic Portosystemic Shunt (TIPS)

SUMMARY:
Creation of the parenchymal tract between the portal vein and the hepatic vein is the most difficult and time consuming step in a TIPS procedure. The purpose of this study is to evaluate portal vein access sets during the TIPS procedure.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of the TIPS procedure
2. TIPS procedure initiated for refractory variceal bleeding, refractory ascites and/or hydrothorax
3. Willing and able to provide written informed consent and HIPAA (Health Insurance Portability and Accountability Act) authorization
4. Willing and able to comply with the study procedures and follow up schedule

Exclusion Criteria:

1. Known active malignancy
2. MELD score ≥ 18 at time of screening
3. History of polycystic liver disease
4. Active bleeding from any source
5. Pulmonary hypertension, heart failure, severe tricuspid valve dysfunction, right to left cardiopulmonary shunt
6. Chronic, occlusive portal vein thrombosis or complete portal vein thrombosis of the main or target portal vein on prior CT examination
7. Active or uncontrolled hepatic encephalopathy
8. Systemic infection/sepsis
9. Biliary obstruction
10. Uncorrectable coagulopathy
11. Any diminutive or partially thrombosed right portal vein
12. Hepatic vein thrombosis (i.e., no Budd-Chiari syndrome)
13. Known sensitivity to contrast or serious contrast reaction such as anaphylaxis
14. Pregnant women or women who are planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Venkatesh P. Krishnasamy, MD, Principal Investigator — New York Presbyterian - Columbia University Medical Center; Danyel C Carr, MS, Study Director — Argon Medical Devices
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - New York Presbyterian - Columbia University Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TIPS With Scorpion Portal Vein Access Kit | TIPS With Cook Transjugular Liver Access Set
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TIPS With Scorpion Portal Vein Access Kit | TIPS With Cook Transjugular Liver Access Set | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Procedural Success
Description: Creation of the parenchymal tract between the hepatic vein and an intrahepatic branch of the portal vein confirmed by portogram (CO2/contrast).
Time Frame: TIPS Procedure (Day 0), up to 93 minutes
Population: 2 participants with Scorpion Portal Vein Access Kit whereas 1 participant with Cook Transjugular Liver Access Set
Measure: Number; unit: Participants
Arm/Group | TIPS With Scorpion Portal Vein Access Kit | TIPS With Cook Transjugular Liver Access Set
Number analyzed (Participants) | 2 | 1
Participants
  Yes | 2 | 1
  No | 0 | 0

2. Primary Outcome: Composite of Major Complications
Description: Major complications associated with the procedure or study device and defined as complications resulting in an unplanned increase in the level of care, prolonged hospitalization, permanent adverse sequelae, or death.
Time Frame: Through 30 days post-TIPS procedure
Measure: Number; unit: Events
Arm/Group | TIPS With Scorpion Portal Vein Access Kit | TIPS With Cook Transjugular Liver Access Set
Number analyzed (Participants) | 2 | 1
Events | 0 | 1

3. Secondary Outcome: Portal Vein Access (PVA) Time
Description: Time (in minutes) from the first forward motion of the needle to confirmation of portal vein access via portogram.
Time Frame: TIPS Procedure (Day 0), up to 52 minutes
Population: 2 participants with Scorpion Portal Vein Access Kit whereas 1 participant with Cook Transjugular Liver Access Set
Measure: Number; unit: minutes
Arm/Group | TIPS With Scorpion Portal Vein Access Kit | TIPS With Cook Transjugular Liver Access Set
Number analyzed (Participants) | 2 | 1
minutes
  Subject ID 02-001: number analyzed (Participants) | 0 | 1
  Subject ID 02-001 |  | 52
  Subject ID 02-002: number analyzed (Participants) | 1 | 0
  Subject ID 02-002 | 7 |
  Subject ID 02-003: number analyzed (Participants) | 1 | 0
  Subject ID 02-003 | 8 |

4. Secondary Outcome: Number of Participants With Technical Success
Description: Creation of a shunt (stent bridging) between the portal and systemic veins.
Time Frame: TIPS Procedure (Day 0), up to 93 minutes
Measure: Number; unit: Participants
Arm/Group | TIPS With Scorpion Portal Vein Access Kit | TIPS With Cook Transjugular Liver Access Set
Number analyzed (Participants) | 2 | 1
Participants
  Yes | 2 | 1
  No | 0 | 0

5. Secondary Outcome: Number of Needle Passes
Description: Count of needle throws between the hepatic and portal vein to create the parenchymal tract.
Time Frame: TIPS Procedure (Day 0), up to 93 minutes
Population: 2 participants with Scorpion Portal Vein Access Kit whereas 1 participant with Cook Transjugular Liver Access Set
Measure: Number; unit: Number of Needle Passes
Arm/Group | TIPS With Scorpion Portal Vein Access Kit | TIPS With Cook Transjugular Liver Access Set
Number analyzed (Participants) | 2 | 1
Number of Needle Passes
  Subject ID 02-001: number analyzed (Participants) | 0 | 1
  Subject ID 02-001 |  | 3
  Subject ID 02-002: number analyzed (Participants) | 1 | 0
  Subject ID 02-002 | 1 |
  Subject ID 02-003: number analyzed (Participants) | 1 | 0
  Subject ID 02-003 | 1 |

6. Secondary Outcome: Procedure Duration
Description: Interval (in minutes) from first jugular access for TIPS creation to removal of catheters from the patient.
Time Frame: TIPS Procedure (Day 0), up to 93 minutes
Population: 2 participants with Scorpion Portal Vein Access Kit whereas 1 participant with Cook Transjugular Liver Access Set
Measure: Number; unit: Minutes
Arm/Group | TIPS With Scorpion Portal Vein Access Kit | TIPS With Cook Transjugular Liver Access Set
Number analyzed (Participants) | 2 | 1
Minutes
  Subject ID 02-001: number analyzed (Participants) | 0 | 1
  Subject ID 02-001 |  | 93
  Subject ID 02-002: number analyzed (Participants) | 1 | 0
  Subject ID 02-002 | 35 |
  Subject ID 02-003: number analyzed (Participants) | 1 | 0
  Subject ID 02-003 | 49 |

7. Secondary Outcome: Fluoroscopy Time
Description: Measured in minutes
Time Frame: TIPS Procedure (Day 0), up to 31.5 minutes
Population: 2 participants with Scorpion Portal Vein Access Kit whereas 1 participant with Cook Transjugular Liver Access Set
Measure: Number; unit: Minutes
Arm/Group | TIPS With Scorpion Portal Vein Access Kit | TIPS With Cook Transjugular Liver Access Set
Number analyzed (Participants) | 2 | 1
Minutes
  Subject ID 02-001: number analyzed (Participants) | 0 | 1
  Subject ID 02-001 |  | 31.5
  Subject ID 02-002: number analyzed (Participants) | 1 | 0
  Subject ID 02-002 | 18.2 |
  Subject ID 02-003: number analyzed (Participants) | 1 | 0
  Subject ID 02-003 | 16.7 |

8. Secondary Outcome: Device-Related Complications
Description: Incidence of complications related to the device as judged by the Investigator
Time Frame: Through 30 days post-TIPS procedure
Population: 2 participants with Scorpion Portal Vein Access Kit whereas 1 participant with Cook Transjugular Liver Access Set
Measure: Number; unit: Number of AEs
Arm/Group | TIPS With Scorpion Portal Vein Access Kit | TIPS With Cook Transjugular Liver Access Set
Number analyzed (Participants) | 2 | 1
Number of AEs
  Subject ID 02-001: number analyzed (Participants) | 0 | 1
  Subject ID 02-001 |  | 2
  Subject ID 02-002: number analyzed (Participants) | 1 | 0
  Subject ID 02-002 | 2 |
  Subject ID 02-003: number analyzed (Participants) | 1 | 0
  Subject ID 02-003 | 4 |

ADVERSE EVENTS:
Time Frame: Adverse event reporting started at the time of the TIPS procedure (on Day 0) and ended at Day 30.
Arm/Group | TIPS With Scorpion Portal Vein Access Kit | TIPS With Cook Transjugular Liver Access Set
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TIPS With Scorpion Portal Vein Access Kit (N=2) | TIPS With Cook Transjugular Liver Access Set (N=1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TIPS With Scorpion Portal Vein Access Kit (N=2) | TIPS With Cook Transjugular Liver Access Set (N=1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Decreased activity (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early due to insufficient enrollment. Three (3) subjects were enrolled before the early termination leading to limited analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT05765253/Prot_SAP_000.pdf